CLINICAL TRIAL: NCT03647566
Title: 18F Sodium Fluoride PET/CT in Acute Aortic Syndrome
Acronym: FAASt
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government); British Heart Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: AC18044
Record Dates: First submitted 2018-04-11; First posted 2018-08-27 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2020-04

CONDITIONS: Acute Aortic Syndrome; Aortic Dissection; Penetrating Aortic Ulcer; Intramural Hematoma
Keywords: sodium fluoride; positron emission tomography; computed tomography; acute aortic syndrome; aortic dissection; intramural haematoma; penetrating aortic ulcer
MeSH Terms: conditions — Acute Aortic Syndrome; Aortic Dissection; Penetrating Atherosclerotic Ulcer | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Aortic tissue specimens obtained from individuals undergoing open surgical repair will be studied histologically, using autoradiography and micro-PET/CT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- No Aortic Disease: Participants with normal calibre aortae and no prior diagnosis of acute aortic syndrome
  Interventions: Diagnostic Test: 18F Sodium Fluoride Positron Emission Tomography / Computed Tomography; Diagnostic Test: Aortic MRI
- Acute Aortic Syndrome: Participants presenting acutely with a diagnosis of acute aortic syndrome as defined in the European Society of Cardiology guidelines: a compatible clinical presentation with CT or magnetic resonance imaging confirming acute aortic syndrome.
  Interventions: Diagnostic Test: 18F Sodium Fluoride Positron Emission Tomography / Computed Tomography; Diagnostic Test: CT Aortic Angiogram
- Chronic Aortic Disease: Participants with an established diagnosis of acute aortic syndrome.
  Interventions: Diagnostic Test: 18F Sodium Fluoride Positron Emission Tomography / Computed Tomography; Diagnostic Test: CT Aortic Angiogram

INTERVENTIONS:
Diagnostic Test: 18F Sodium Fluoride Positron Emission Tomography / Computed Tomography — PET scan using the 18F-Sodium Fluoride radiotracer followed by an attenuation correction CT scan
Diagnostic Test: CT Aortic Angiogram — CT scan to assess aortic morphology and contextualise PET scan
  Groups: Acute Aortic Syndrome; Chronic Aortic Disease
Diagnostic Test: Aortic MRI — Aortic MRI to assess aortic morphology and contextualise PET scan
  Groups: No Aortic Disease

SUMMARY:
The purpose of this study is to determine whether Sodium Fluoride imaging (using Positron Emission Tomography-Computed Tomography - PET-CT) is able to predict disease progression in acute aortic syndrome.

DETAILED DESCRIPTION:
Acute Aortic Syndrome encompasses multiple aortopathies, including aortic dissection, intramural haematoma and penetrating aortic ulcers. Acute aortic syndrome has a three year mortality approaching 25%. To date, other than the initial aortic diameter, there are no accurate methods of establishing the risk of disease progression in patients with acute aortic syndrome.

In vascular disease, microcalcification occurs in response to necrotic inflammation. Using computed tomography and positron emission tomography (PET-CT), early microcalcification can be identified using uptake of the radiotracer 18F-sodium fluoride. This can identify high risk-lesions in the aorta, coronary and carotid arteries, and appears to be indicative of necrotic and heavily inflamed tissue. In abdominal aortic aneurysms, 18F-sodium fluoride binding predicts aortic expansion and the risk of aneurysm rupture or requirement for surgical repair.

The study investigators, therefore, propose to evaluate the ability of 18F-sodium fluoride to identify regions of necrotic inflammation in acute aortic syndrome to predict aortic expansion and disease progression.

Control patients with a normal calibre aorta will be recruited from the National Abdominal Aortic Aneurysm Screening Programme and Vascular Out-Patient Clinics. Patients with acute aortic syndrome and chronic aortic disease will undergo clinical assessments and 18F Sodium Fluoride PET/CT scans at baseline and 12-months. Clinical follow-up will continue for up to 3 years from recruitment.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients with Acute Aortic Syndrome or Chronic Aortic Disease:

* A diagnosis of acute aortic syndrome as defined as per the European Society of Cardiology guidelines on the management of aortic disease a compatible clinical presentation with CT or magnetic resonance imaging confirming acute aortic syndrome.
* Adults over the age of 25 years
* Participants who have had previous open or thoracic endovascular aortic repair (TEVAR) are eligible to participate in the study.

Healthy Controls:

* No previous diagnosis of aortic disease
* Over the age of 55 years

EXCLUSION CRITERIA:

* The inability of patients to undergo PET/CT scanning
* Chronic kidney disease (eGFR ≤ 30 mL/min/1.73 m2)
* Major or untreated cancer
* Pregnancy
* Allergy or contra-indication to iodinated contrast
* Inability or unwillingness to give informed consent

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with acute aortic syndrome will be recruited from emergency hospital admissions. Participants with chronic aortic disease will be recruited from out-patient clinics and thoracic aortic surveillance programmes. Healthy volunteers will be recruited from the national abdominal aortic aneurysm screening service and vascular out-patient department clinics.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Aortic diameter | 12 months
  Maximum cross-sectional aortic diameter

SECONDARY OUTCOMES:
18F Sodium Fluoride uptake in the aorta | 12 months
  18F Sodium Fluoride binding in the aorta will be measured from PET/CT scans performed at recruitment and at 12 months follow-up. Uptake will be quantified in Standardised Uptake Values and as a tissue to background ratios.
Hospital admissions | 24 months
  The requirement for hospital admission
Surgical Intervention | 24 months
  Requirement for surgical intervention during follow-up period
Change in renal function | 24 months
  Creatinine change during the follow-up period
Short Form-12 (SF12) questionnaire score | 24 months
  The SF12 is a validated, self reported quality of life assessment questionnaire. It consists of 12 questions that measure functional and mental well-being. Scores range from 12 to 47.
Disease related survival | 24 months
  Disease related survival
All-cause mortality | 24 months
  All-cause mortality

OTHER OUTCOMES:
Co-localisation of 18F-Sodium Fluoride with histological changes in aortic tissue | 12 to 36 months
  Uptake of 18F-Sodium Fluoride will be identified on PET-CT scans that are acquired as part of the study visit. This will be compared with histological changes in aortic specimens obtained from participants undergoing open surgical repair.

CONTACTS AND LOCATIONS:
Overall Officials: Maaz BJ Syed, MBChB MSc, Principal Investigator — University of Edinburgh
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared outside the current research group

REFERENCES:
- [Derived] Syed MBJ, Fletcher AJ, Debono S, Forsythe RO, Williams MC, Dweck MR, Shah ASV, Macaskill MG, Tavares A, Denvir MA, Lim K, Wallace WA, Kaczynski J, Clark T, Sellers SL, Masson N, Falah O, Chalmers RTA, Tambyraja AL, van Beek EJR, Newby DE. 18F-Sodium Fluoride Positron Emission Tomography and Computed Tomography in Acute Aortic Syndrome. JACC Cardiovasc Imaging. 2022 Jul;15(7):1291-1304. doi: 10.1016/j.jcmg.2022.01.003. Epub 2022 Mar 16. PMID 35798405